CLINICAL TRIAL: NCT04513769
Title: Nutritious Eating With Soul at Rare Variety Cafe: Local Dissemination and Implementation
Brief Title: Nutritious Eating With Soul at Rare Variety Cafe
Acronym: NEWSoul@RV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, John Bernhart, Principal Investigator, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100991
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): This is a single-arm study so all participants receive the same intervention.
  Interventions: Behavioral: Vegan diet

INTERVENTIONS:
Behavioral: Vegan diet — Participants will receive a behavioral intervention on a vegan diet in partnership with a local vegan soul food restaurant

SUMMARY:
To date, few dissemination and implementation (D&I) studies exist of successful healthy eating interventions delivered through restaurant settings. Therefore, the proposed study will investigate the following aims:

Aim 1: Examine reach and adoption of a modified, 12-week NEW Soul vegan intervention delivered through a train-the-trainer approach in a soul food vegan restaurant.

Aim 2: Assess resource use and cost associated with a train-the-trainer D&I approach in a restaurant setting.

Aim 3: Examine effectiveness through changes in participants' diet, self-efficacy, weight loss, and quality of life from baseline to follow-up (3-months) and at maintenance (9-months).

Aim 4: Assess implementation fidelity and participant satisfaction of modified NEW Soul.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American
* between 18-65 years old
* be free on meeting night (Tuesday at 6PM)
* be free of eating disorder
* be free of major health or psychiatric diseases, drug or alcohol dependency, thyroid conditions, diabetes, or pregnancy
* willing to travel weekly to Rare Variety Café

Exclusion Criteria:

* currently following a plant-based/vegan diet
* have a body mass index of under 25 or over 49.9 kg/m2
* currently on medication for diabetes
* women who are currently pregnant or breastfeeding (or plan to become pregnant in the next 24 months)
* currently participating in a weight loss program or taking weight loss medications
* recent weight loss (>10lbs in the last 6 months)
* living in the same household as somebody already participating in the larger NEW Soul Study at the University of South Carolina
* currently in the NEW Soul study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
body weight | 0, 3, and 12 months
  Assess changes in body weight

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernhart JA, Turner-McGrievy GM, Wilson MJ, Sentman C, Wilcox S, Rudisill C. NEW Soul in the neighborhood-reach and effectiveness of a dissemination and implementation feasibility study. Transl Behav Med. 2023 Apr 3;13(3):123-131. doi: 10.1093/tbm/ibac080. PMID 36689305